CLINICAL TRIAL: NCT00747370
Title: The Suitability of Dynamic MRI for Pelvic Floor, Bladder Neck and Midurethra
Brief Title: Dynamic MRI of the Behaviour of Female Pelvic Floor
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Kirsi Rinne, Kuopio University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: KUH5302421
Record Dates: First submitted 2008-09-03; First posted 2008-09-05 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-09

CONDITIONS: Stress Urinary Incontinence; Genital Prolapse
Keywords: stress urinary incontinence; Tension free vaginal tape; tension free vaginal tape obturator; genital prolapse
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other): 16 healthy volunteers with no complaints of urinary symptoms and without urogenital prolapse of more than first degree.
  Interventions: Procedure: movement of midurethra, bladder neck, cervix and rectum
- 2 (Other): Forty two stress urinary incontinence patients without prior urogenital prolapse or incontinence operation and without genital prolapse more than first degree
  Interventions: Procedure: movement of midurethra, bladder neck, cervix and rectum
- 3 (Other): 16 genital prolapse women without prior prolapse operations or any symptoms of incontinence
  Interventions: Procedure: movement of midurethra, bladder neck, cervix and rectum

INTERVENTIONS:
Procedure: movement of midurethra, bladder neck, cervix and rectum

SUMMARY:
The purpose of this study was to test the suitability of dynamic magnetic resonance imaging for the pelvic floor floor, bladder neck and urethra in healthy volunteers, in stress incontinent patient and in women with genital prolapse.

DETAILED DESCRIPTION:
Traditional methods for evaluation of urinary incontinence in women include urodynamics, cystourethroscopy, cystourethrography and ultrasonography.Magnetic resonance imaging (MRI) offers a new tool for evaluation of morphology and function of the urogenital compartment of the female pelvis. Moreover, MRI gives opportunity to study function of the pelvic floor organs in terms of mobility and reactions during different physiological and provocative activities.

The aim of the present study was by means of dynamic MRI to evaluate the behaviour of the mid-urethra, bladder neck, cervix and rectum in different maneuvers in three different study groups. Sixteen healthy volunteers with no complaints of urinary symptoms or urogenital prolapses, 42 stress urinary incontinence patients and 16 women with third degree genital prolapse were examined respectively.

ELIGIBILITY:
Inclusion Criteria:

* healthy women without any urogenital symptoms
* stress urinary incontinence ( group II )
* genital prolapse of third degree ( group III)

Exclusion Criteria:

* previous incontinence or prolapse surgery
* lower urinary tract anomaly
* current UTI or > 3 UTI episodes within the past year
* previous radiation therapy of the pelvis
* active malignancy
* neurogenic disease which can be associated with bladder disorders
* patient unable to understand the purpose of the study
* patient immobile

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2002-01; Primary Completion 2007-12 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The movement of midurethra, bladder neck, cervix and rectum measured by dynamic MRI | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gynecology and Radiology, Kuopio University Hospital, Kuopio, Finland